CLINICAL TRIAL: NCT07179107
Title: Adequate Hydration and Health Outcomes
Acronym: HYDRATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FP00043890
Record Dates: First submitted 2025-09-04; First posted 2025-09-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dehydration; Dehydration (Physiology); Glucose Abnormalities; Cardiovascular
Keywords: hydration; dehydration; underhydration; fluid intake; non caloric sweeteners
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial. Data collection will cover a period of 3 years.
  Each participant will be part of the study for 8 weeks. Each testing day, once a week will last 3.5 hours. First subject in September 2025 and last subject out July 2028
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Baseline - week 1 (Other): Habitual fluid intake during week 1 of the study
  Interventions: Other: Baseline - week 1
- Low Water intake - week 2 (Experimental): Low water intake as described by the protocol
  Interventions: Other: Low Water Intake - week 2
- Moderate water intake - week 3 (Experimental): Moderate water intake as described by the protocol
  Interventions: Other: Moderate Water Intake - week 3
- Adequate Water intake - Week 4 (Experimental): Adequate water intake as described by the protocol
  Interventions: Other: Adequate Water Intake - week 4
- Washout period - week 5 (Other): Habitual fluid intake week
  Interventions: Other: Washout - week 5
- Low fluid intake with non caloric sweeteners - Week 6 (Experimental): Low fluid intake with non-caloric sweeteners - Week 6
  Interventions: Other: Low fluid intake with non caloric sweeteners - Week 6
- Moderate fluid intake with non caloric sweeteners - Week 7 (Experimental): Moderate fluid intake with non caloric sweeteners - Week 7
  Interventions: Other: Moderate fluid intake with non caloric sweeteners - Week 7
- Adequate fluid intake with non caloric sweeteners - Week 8 (Experimental): Adequate fluid intake with non caloric sweeteners - Week 8
  Interventions: Other: Adequate fluid intake with non caloric sweeteners - Week 8

INTERVENTIONS:
Other: Baseline - week 1 — Habitual fluid intake during week 1
  Arms: Baseline - week 1
Other: Low Water Intake - week 2 — Low water intake as described by the protocol
  Arms: Low Water intake - week 2
Other: Moderate Water Intake - week 3 — Moderate Water Intake - Week 3
  Arms: Moderate water intake - week 3
Other: Adequate Water Intake - week 4 — Adequate Water Intake - week 4
  Arms: Adequate Water intake - Week 4
Other: Washout - week 5 — Washout - week 5
  Arms: Washout period - week 5
Other: Low fluid intake with non caloric sweeteners - Week 6 — Low fluid intake with non caloric sweeteners - Week 6
  Arms: Low fluid intake with non caloric sweeteners - Week 6
Other: Moderate fluid intake with non caloric sweeteners - Week 7 — Moderate fluid intake with non caloric sweeteners - Week 7
  Arms: Moderate fluid intake with non caloric sweeteners - Week 7
Other: Adequate fluid intake with non caloric sweeteners - Week 8 — Adequate fluid intake with non caloric sweeteners - Week 8
  Arms: Adequate fluid intake with non caloric sweeteners - Week 8

SUMMARY:
Cardiovascular diseases (CVD) are the leading cause of death in middle- and high-income countries, according to data from the World Health Organization (WHO). Epidemiological studies have associated low water intake and underhydration with diabetes, chronic kidney disease, and an increased risk of CVD. Similarly, the prevalence of chronic metabolic dysfunction is increasing dramatically worldwide, becoming both a significant public health concern and a global economic burden. Reports from the WHO indicate that the number of people with diabetes worldwide has risen from 108 million in 1980 to 422 million in 2014, representing 8.5% of adults. Therefore, there is an urgent need to identify modifiable risk factors that could help prevent metabolic dysfunction and mitigate the epidemic of type 2 diabetes (T2D). Evidence suggests that the hormone arginine vasopressin (AVP) may play a key role. AVP is the primary hormone responsible for regulating body fluid balance; however, increased AVP secretion, such as under conditions of low water intake, appears to be a risk factor for developing diabetes.

Increasing water intake may represent a simple and cost-effective way to improve glucose regulation and cardiovascular health. However, many individuals do not prefer drinking plain water, and although beverages with high sugar content may promote greater fluid intake, they also contribute additional calories that can negatively impact body weight and overall health. Thus, the central research question of this study is whether improving hydration with non-sugar-sweetened beverages can provide equivalent benefits for hydration and health outcomes in adults.

Aim 1: To explore the association between habitual fluid intake and fluid preferences (water and non-sugar-sweetened beverages), hydration biomarkers, and health outcomes in normal-weight and obese adults.

Aim 2: To compare the impact of increased total water intake, provided as plain water or non-sugar-sweetened beverages, on hydration, cardiovascular health, and glucose regulation in normal-weight and obese adults.

DETAILED DESCRIPTION:
Protocol

Subjects will first come into the lab for a screening visit (approximately 1 hour). In this visit, they will learn more about the study, provide written informed consent (if they choose to participate), fill out a medical history form, have their weight, height, and body composition measured, and have a finger stick blood test to measure glycosylated hemoglobin (HbA1c). Those with A1c values >7% at screening will not be included in the study. We will provide them with information about HbA1c levels that meet the diagnostic criterion for diabetes immediately. Those with A1c values from 6.5 to ≤7% will be provided with information about HbA1c levels that meet the diagnostic criterion for diabetes at the end of the trial. We will suggest they share this information with their doctor. We will answer any questions they may have.

Two groups of 72 volunteers each will be grouped as having normal weight or obesity based on their BMI. The subjects who enroll in the study will undergo an 8-week cross-ver study with two separate arms based on BMI category. Subjects in each BMI category will be evaluated weekly as described below and depicted in Figure 1:

Week 1: Baseline. During this week, the subjects will maintain their habitual fluid intake without any intervention.

Weeks 2-4 & Weeks 6-8: All subjects will follow 3 weeks of consuming only plain water and a 3-week of non-sugar sweetened beverages, in a random order.

Weeks 2 and 6: The subject will consume very-low fluid intake, of 1.2 and 1.5 L/day for females and males, respectively.

Week 3 & week 7: Subjects will consume low fluid intake, of 1.6 and 2.0 L/day for females and males, respectively.

Week 4 & week 8: Subjects will consume adequate fluid intake according to the US dietary guidelines (2.2 and 3.0 L/day L/day for females and males, respectively).

Week 5: Wash-out period, where subjects can return to their habitual fluid and dietary intake.

Fluid intake:

Fluid intake will be controlled by providing drinks and programmable smart water bottles to record ﬂuid intake and provide periodic reminders.

Plain Water:

During the 3 weeks, subjects will be instructed to consume ﬂuids only in the form of plain water (tap, bottle, sparkling), coffee up to 1 cup a day, and alcohol, up to 2 servings per week only during week 5 but not anywhere else during the study.

Non-Sugar-Sweetened beverages:

During the 3-week period, of the NSSB portion of the study 1.0 L of ﬂuids per day will be coming from non-sugar-sweetened beverages, with the rest coming from water.

Procedures:

During this study, beverages will be provided for participants. Programmable smart water bottles will be used to record fluid intake and provide periodic reminders.

Participants will be instructed to keep their diet as usual, without making any changes during the study. The ASA24 will be administered at the end of weeks 1, 2, 3, 4, 5, 6, 7, and 8. The volunteers will be asked to fill out 24-hour recalls (ASA24) three times each one of the weeks 1, 2 and 3. We will collect 2 weekdays and 1 weekend day. ASA24 is an online nutritional assessment tool developed by the NCI.

1 Week before data collection begins: Subjects will visit the lab to place the CGM for baseline data collection, distribute frozen meals, watches, urine containers, and water bottles.

Day Before each Testing:

During the 24 hours prior to each testing day, subjects will be provided with verbal and written instructions on the 24-h urine collection protocol and two 3L urine collection containers, which will include the preservative. They will be asked to collect all their urine beginning with the second void of the day. The first morning urine sample will not be collected; the second void on the day before testing will begin the 24-hour collection. The last urine sample to be collected will be the first morning urine sample of the testing day in a separate container. To measure compliance with the 24-h urine collection protocol, subjects will be asked to complete a 24-h urine collection log. They will record the time when they collect the urine samples, and if they missed any voids. Urine will be analyzed for hydration measures, urine creatinine, and non-nutritive sweeteners. Also participants will have to consume the same dinner before each one of the 8 lab visits, that will be provided in the form of frozen meal from the research team.

TESTING DAYS Each subject will visit the lab once a week for 8 consecutive weeks after at least 10 h of fasting. Upon arrival in the lab, subjects will provide a urine sample measured for hydration biomarkers and their body weight and body composition will be assessed on a bioelectrical impedance scale. We will acess seated blood pressure. Next, participants will fill out cognitive and perceptual questionaires. After this we will access resting metabolic rate, endothelial function by flow mediated dilation (FMD). After the completion of the FMD test, we will proceed to the oral glucose tolerance test (OGTT).

Glycemic Test:

Three separate glycemic tests will be performed depending on the stage of the protocol:

1. Insulin Resistance on Matthews's homeostatic model assessment of insulin resistance (HOMA-IR) is based on fasting glucose and insulin.
2. Oral Glucose Tolerance Test (OGTT). This 120-minute test consists of a fasted blood sample followed by 75 grams of glucose solution ingestion. Four more blood samples will be collected 30, 60, 90, and 120 minutes after the ingestion.
3. Ambulatory 24-hour glucose responses will be assessed via continuous glucose monitor (CGM) during the 7-week intervention. Each CGM lasts for 14 days, thus 4 monitors will be used for each volunteer. The Abbott libre pro will be used to asses interstitial blood glucose every 15 min.

Blood Analysis:

Fasting blood samples will analyzed for :

* Glucose and insulin to assess insulin resistance based on Matthews's homeostatic model assessment of insulin resistance (HOMA-IR).
* Osmolality, sodium, and copeptin for hydration assessment.
* Glucagon and cortisol, since both are stimulated by vasopressin, and impacting glucose regulation.

Blood Samples during the Oral Glucose Tolerance Test (OGTT) will be analyzed:

- Glucose, insulin, glucagon, and cortisol. The primary outcome of the OGTT will be the area under the curve for glucose, insulin, glucagon, and cortisol during the 120-minute test.

Cognitive Data:

A neuropsychological test measuring such aspects of cognition as attention, executive function and memory will be administered to each subject. We will ask participants to complete a cognitive task designed to examine mostly their Executive function (inhibition) abilities, named the Flanker's test. The task will be administered on a laptop computer, lasts 5 minutes and will be given at each visit.

Perceptual Data:

Perceptual data on hunger, cravings, thirst, and mouth dryness will be collected in a pen and paper format.

Mood Assessment:

Mood will be assessed by the validated thirty-five-question Adult Short Profile of Mood States (POMS) questionnaire (POMS 2®-A Short, Multi-Health Systems Inc.). It will be administed on a laptop computer and it lasts 5 min

Sleep Quality Assessment:

This will be assessed via the Pittsburgh Sleep Quality Index. This is a short questionnaire that takes about 2-3 minutes to fill out. The sleep quality assessment will be completed on paper.

Resting Blood pressure:

After the cognitive/ perceptual test, a resting blood pressure in seated position will be taken with and automated blood pressure cuff in duplicate.

Resting Metabolic Rate:

Resting metabolic rate via indirect calorimetry for 30 minutes. This will take place while subjects are resting prior to the flow mediated dilation test.

Flow Mediated Dilation Test:

Endothelium-dependent, FMD of the brachial artery is assessed at baseline (pre-condition) and at the end of each visit (post-condition), at the end of weeks 1, 2, 3, 4, 5, 6, 7, and 8. Measurement procedures are done in accordance with established guidelines and performed by a registered sonographer using B-mode ultrasound (Philips Epic Elite™,Bothell WA). FMD analyses are conducted in a dim, quiet, temperature-controlled environment (22-25 oC) with the participants lying down on an ultrasound bed. Participants will be sized for appropriate blood pressure cuff (Hokanson Instruments, Bellevue, WA) and cuff will be placed around the right arm, 2-3 cm below the elbow/forearm area. Simultaneous ultrasound images (B-mode) and doppler waveforms of the brachial artery are captured for baseline before the blood pressure cuff is inflated to a suprasystolic pressure of 250 mmHg for 5 minutes. After 5 minutes, the cuff will be rapidly deflated, and arterial images will be obtained for 6 minutes post-inflation. Subjects may experience mild discomfort as the cuff is inflated on the upper arm. The images are obtained and analyzed by a trained, blinded researcher using an automated, previously validated FMD software.

Oral Glucose Tolerance Test (OGTT):

Before this test, an indwelling catheter will be placed in an antecubital vein by a trained and experienced phlebotomist using sterile techniques. After a couple of minutes of rest, a baseline blood sample will be taken and the subject will ingest a drink containing 75 g glucose. Four more blocatheterd samples will be taken at 30, 60, 90, and 120 minutes after the drink ingestion. Blood samples will be analyzed for glucose, insulin, glucagon, cortisol, and copeptin. Extra plasma and serum aliquots will be stoford in the deep freezer to -nalysis of other health related biomarkers. The first blood sample will be 15 mL and the remaining four samples will be 10 mL. The total volume for each test will be 55 mL.The total blood volume for all samples during the eight testing sessions will be 440 mL, which is equivalent to a blood donation.

Continuous Glucose Monitor (CGM):

Ambulatory glucose measurements will be obtained using CGM sensors during the entire 8-week period. Since the sensors work for 14 days, a new sensor will be used every two weeks and placed on an alternate arm. The Abbot FreeStyle Libre Pro sensor will be used and it will be applied at the back of the upper arm. A protective round band-aid will also be used to ensure the sensor will not fall off.

Physical Activity:

Physical activity will be assessed via the validated International Physical Activity Questionnaire (IPAQ). This questionnaire will take approximately 2 minutes to complete. Participants will take the questionnaire on paper. The questionnaire will be administered at the end of weeks 1, 2, 3, 4, 5, 6, 7, and 8. IPAQ data will be expressed as a continuous variable of MET-min per week and a three-level categorical variable of physical activity level.

Also, participants will wear a Garmin smart watch that provides heart rate, sleep quality, and time spent on different levels of physical activity. Participants will wear this watch for the entire duration of the intervention. Researchers will provide the watch, and participants will be required to return the watch upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-24.9 or 30.0-39.9 kg/m2
* HbA1c ≤7%
* Age 20-65 y
* available for 8 consecutive weeks same day and time

Exclusion Criteria:

* Diabetes
* HbA1c >7% BMI ≤18.5, BMI of 25 to <30, or ≥ 40 kg/m2
* night shifting work
* losing or gaining weight during the last 2 months (>5 lbs. fluctuation)
* thyroid medication
* bariatric surgery
* Habitual strenuous exercise (>120 min/week) Strenuous exercise is defined as activities that take hard physical effort and make you breathe much harder than normal.
* Construction and other workers that spend signifant portion of their work day outdoors
* Commuting by bicycle
* Eating disorders
* Use of aspirin during the duration of the study
* Cancer
* Renal disease (including kidney stones or recurrent urinary track infections
* Hepatic disease
* Cardiac conditions
* Current infection requiring medication
* Chronic, contagious, infectious diseases such as tuberculosis, Hepatitis A, B, C, or HIV
* Medication that could affect appetite or body weight regulation
* GLP1-RA medication
* Anti-depressent SSRI medication
* Testosterone replacement therapy
* Participating in another study at the same time
* Unable to abstain from alcohol during the study
* Unable to limit caffeinated beverage intake to 1 cup per day
* Donated blood during the past two months
* Uneasibly acessable veins
* Does not have smart phone

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-07-02 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation % | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Flow-mediated dilation (FMD) will be assessed as a non-invasive measure of endothelial function using brachial artery ultrasound. A high-resolution ultrasound probe will measure baseline artery diameter, then artery diameter after 5 minutes of forearm cuff occlusion, followed by rapid cuff deflation. FMD% will be calculated as a percent of [(Maximum Post-Deflation Diameter - Baseline Diameter)/Baseline Diameter]×100 This outcome provides the percent increase in brachial artery diameter relative to baseline, reflecting endothelium-dependent vasodilation.
Area under the curve for glucose | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  The positive integer of the glucose levels during the 120 minutes post ingestion of 75 g of glucose
Insulin area under the curve | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  The positive integer of the insulin levels during the 120 minutes post ingestion of 75 g of glucose
glucagon area under the curve | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  The positive integer of the glucagon levels during the 120 minutes post ingestion of 75 g of glucose
Cortisol area under the curve | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  The positive integer of the cortisol levels during the 120 minutes post ingestion of 75 g of glucose
Mean glucose | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Mean weekly interstitial glucose from the continuous glucose monitor
Glycemic Variability | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  coefficent of variation (%) of weekly interstitial glucose from the continuous glucose monitor
Serum copeptin | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Serum copeptin/vasopressin at baseline of the oral glucose tolerance test
Plasma Sodium | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Plasma sodium at baseline of the oral glucose tolerance test
Plasma Osmolality | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Plasma osmolality at baseline of the oral glucose tolerance test
Total Water Intake | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Weekly average total water intake from Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Urine volume | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  24 hours urine volume the day prior to the oral glucose tolerance test
Urine Osmolality | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Urine Osmolality from a 24 hours urine sample the day prior to the oral glucose tolerance test
Reaction time | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Reaction time assessed via Erikson Flankers Test
Accuracy of cognitive test | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Accuracy on the Erikson Flankers cognitive test
Homeostasis Model Assessment of Insulin Resistance | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention based on the baseline (0 minutes) fasting blood sample.
  The Homeostasis Model Assessment of Insulin Resistance (HOMA-IR), as described by Matthews et al., is a validated index used to estimate insulin resistance from fasting plasma glucose and insulin concentrations. It is commonly applied in clinical trials as a practical and reliable surrogate measure of insulin sensitivity when clamp techniques are not feasible.

SECONDARY OUTCOMES:
Confusion-bewilderment | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Confusion-bewilderment assessment via the short version of Profile of Mood State Questionnaire. Score range 0-20 with higher score indicating negative mood descriptor
Depression-dejection | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Depression-dejection assessment via the short version of Profile of Mood State Questionnaire. Score range 0-20 with higher score indicating negative mood descriptor
Fatigue-inertia | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Fatigue-inertia assessment via the short version of the Profile of Mood State Questionnaire. Score range 0-20, with higher score indicating a negative mood descriptor
Vigour-activity | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Vigour-activity assessment via the short version of Profile of Mood State Questionnaire. Score range 0-20 with higher score indicating positive mood descriptor
Total mood disturbance | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Total mood disturbance assessment via the short version of the Profile of Mood State Questionnaire. Score range 0-120, with higher score indicating overall negative mood descriptor
Thirst | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Thirst assessed via a visual analog scale
Hunger | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Hunger assessed via a Visual Analog scale
Total Body Water | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Total Body Water assessed via SOZO multiple frequency bioelectrical impedance spectroscopy
Intracellular Water | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Intracellular Water assessed via SOZO multiple frequency bioelectrical impedance spectroscopy
Extra cellular water | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Extra cellular water assessed via SOZO multiple frequency bioelectrical impedance spectroscopy
Cravings | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Cravings assessed via a five questions with a score out of 25
Urine acesulfame potassium | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Urine acesulfame potassium assessed from 24 urine sample the day prior to the oral glucose tolerance test
Urine Sucralose | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Urine sucralose assessed from 24 urine sample the day prior to the oral glucose tolerance test
Resting Energy Expenditure | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Resting Energy expenditure assessed by indirect calorimetry with canopy
Resting Energy expediture from fat oxidation | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Resting Energy expediture from fat oxidation assessed by indirect calorimetry with canopy
Resting energy expenditure from carbohydrates oxidation | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Resting energy expenditure from carbohydrates oxidation assessed by indirect calorimetry with canopy
Total Caloric Intake | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Total Caloric intake from Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Total Sodium intake | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Total Sodium intake assessed by the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool
Total Protein intake | 1, 2, 3, 4, 5, 6, 7, 8 weeks of the intervention
  Total Protein Intake from the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - 850 PBC, Phoenix, Arizona
  - 850 Phoenix Bioscience Core, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No